CLINICAL TRIAL: NCT05822531
Title: Promoting Cardiovascular Health of Northern Appalachian Women During and After Pregnancy: PSU Maternal Pilot Study
Brief Title: Early Intervention to Promote Cardiovascular Health of Mothers and Children (ENRICH) During Pregnancy
Acronym: ENRICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ian M. Paul, M.D., M.Sc., Professor of Pediatrics and Public Health Sciences; Chief, Division of Academic General Pediatrics; Vice Chair of Faculty Affairs, Department of Pediatrics Affiliation: Penn State University, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00021577; 1UG3HL162971-01 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-20 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Pregnancy Related; Sedentary Behavior
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This pilot study is being conducted to inform feasibility of the next phase of this research project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maternal Cardiovascular health (CVH) Intervention (Experimental): The pilot maternal CVH intervention will be delivered by NFP partners starting as early as NFP program enrollment in the first trimester after confirmation of a viable pregnancy and no later than the 28th week of pregnancy and will continue up to 6 months postpartum. The visit schedule will be consistent with the NFP visit structure to deliver intervention content at regularly scheduled visits that are typically 60 minutes long (weekly visits for the first month following enrollment followed by twice monthly visits until delivery). The pilot study will include an enhanced behavioral component target decreased sedentary time and increase physical activity and utilizing a technology/monitoring component. All women be monitored using a wrist-worn actigraphy device to record daily activity, intermittent home blood pressure self-monitoring, intermittent home weight self-monitoring, and carbon monoxide monitoring administered by the NFP nurse.
  Interventions: Behavioral: Maternal CVH Intervention

INTERVENTIONS:
Behavioral: Maternal CVH Intervention — All participants will be enrolled into the intervention arm of this pilot study.

SUMMARY:
This pilot study aims to examine the feasibility and acceptability of adding a cardiovascular health module to the existing Nurse Family Partnership (NFP) home visitation program delivered by trained nurses in the Northern Appalachian region of Central Pennsylvania.

DETAILED DESCRIPTION:
The Promoting Cardiovascular Health of Northern Appalachian Women During and After Pregnancy: Pilot Study is a single arm pilot study that will enroll pregnant women (<28 weeks' gestation) participating in the NFP home visitation program in the Northern Appalachian region of Central Pennsylvania. This pilot study will include an enhanced version of the NFP standard care plan delivered by trained nurses to promote cardiovascular health among women by targeting decreased sedentary time and enhanced physical activity (and where applicable smoking cessation) during and after pregnancy. This pilot study will also examine the feasibility and acceptability of digital devices (actigraphy, digital scale, blood pressure monitor) during this same time period.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous pregnant woman
2. Age ≥ 18 years old
3. Enrolled in and receiving the Nurse-Family Partnership program through the Geisinger Clinic or UPMC Home Health Care of Central PA
4. English speaking
5. Women with a singleton viable pregnancy confirmed by NFP home visitors
6. Access to reliable internet service required for data collection
7. A minimum of 5 women with use of nicotine containing products (cigarette, cigar, hookah, chewing tobacco, e-cigarette, patch) within the past 3 months

Exclusion Criteria:

1. Unable or unwilling to comply with the study visits and procedures
2. Participation in a concurrent interventional study
3. Diagnosis of cancer
4. A personal history of complex congenital heart disease
5. A fetus in the current pregnancy with known chromosomal abnormalities or birth defects inconsistent with survival to 2 years will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Women
Enrollment: 12 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, MSc, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - UPMC Home Health, Altoona, Pennsylvania
  - Geisinger, Danville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Maternal Cardiovascular Health (CVH) Intervention
Started | 12
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Maternal Cardiovascular Health (CVH) Intervention
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Integrating a Cardiovascular Health Module to the Existing Nurse-Family Partnership (NFP) Home Visiting Program as Measured by Qualitative Feedback From Home Visitors.
Description: Feasibility will be determined good acceptability by NFP nurses as assessed qualitatively during group discussions. Nurses will use their experience as home visitors to provide feedback to study personnel on whether they are able to successfully integrate new visit content into their usual workflow. They will further give suggestions for future improvement after completion of this pilot study.
Time Frame: 6 months
Population: Qualitative feedback from nurses
Measure: Number; unit: Participants reporting success
Arm/Group | Maternal Cardiovascular Health (CVH) Intervention
Number analyzed (Participants) | 7
Participants reporting success | 7

ADVERSE EVENTS:
Time Frame: Enrollment during pregnancy until 6 months postpartum (up to 12 months)
Groups:
- Pregnancy Loss: cardiovascular health intervention
Arm/Group | Pregnancy Loss
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT05822531/Prot_SAP_ICF_000.pdf